CLINICAL TRIAL: NCT03197298
Title: Clopidogrel or Ticagrelor in Acute Coronary Syndrome Patients Treated With Newer-Generation Drug-Eluting Stents: CHANGE DAPT
Brief Title: Change of Dual Antiplatelet Therapy in Patients With Acute Coronary Syndrome
Acronym: CHANGE DAPT
Status: Completed | Type: Observational
Sponsor: Thorax Centrum Twente (Other)
Responsible Party: Sponsor
Other Study IDs: K14-22
Record Dates: First submitted 2017-05-23; First posted 2017-06-23 (Actual); Last update posted 2017-06-23 (Actual); Status verified 2017-06

CONDITIONS: Acute Coronary Syndrome; Percutaneous Coronary Intervention; Drug-Eluting Stents
Keywords: Acute Coronary Syndrome; Percutaneous Coronary Intervention; Drug-Eluting Stents; Platelet Aggregation Inhibitors; Ticagrelor; clopidogrel; Purinergic P2Y Receptor Antagonists
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Clopidogrel; Ticagrelor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year

GROUPS / COHORTS (2):
- Clopidogrel Period: ACS patients treated by PCI with newer-generation DES before the guideline suggested change in primary DAPT-regimen
  Interventions: Drug: Clopidogrel
- Ticagrelor Period: ACS patients treated by PCI with newer-generation DES after the guideline suggested change in primary DAPT-regimen
  Interventions: Drug: Ticagrelor

INTERVENTIONS:
Drug: Clopidogrel
  Other Names: Plavix
  Groups: Clopidogrel Period
Drug: Ticagrelor
  Other Names: Brilinta; Brilique
  Groups: Ticagrelor Period

SUMMARY:
Acute coronary syndrome (ACS) guidelines have been changed, favoring dual antiplatelet therapy (DAPT) with the more potent P2Y12 inhibitor ticagrelor over clopidogrel (besides aspirin). This change is based on studies that showed benefits of ticagrelor. However, study participants were only partly treated by percutaneous coronary intervention (PCI). In patients who were treated by PCI, this was generally performed using of bare metal or first-generation drug-eluting stents (DES).

CHANGE DAPT is an investigator-initiated, prospective, single centre registry, in which we evaluate the impact of the guideline suggested change in the primary DAPT regimen (from clopidogrel to ticagrelor) on 1-year clinical outcome in ACS patients treated by PCI with newer-generation DES in the Thoraxcentrum Twente.

ELIGIBILITY:
Inclusion Criteria:

* Presentation with acute coronary syndrome (ACS)
* Treated with newer-generation drug-eluting stent (DES) in coronary artery or bypass graft lesion

Exclusion Criteria:

* Known pregnancy
* Life expectancy less than one year
* Planned elective surgery requiring interruption of DAPT in the first 6 months
* Known intolerance to components of the DES available
* Indication for oral anticoagulation at baseline

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the primary cardiac care clinic of the Thoraxcentrum Twente
Sampling Method: Probability Sample
Enrollment: 2062 (Actual)
Dates: Start 2012-12-21 (Actual); Primary Completion 2016-07-25 (Actual); Study Completion 2016-07-25 (Actual)

PRIMARY OUTCOMES:
Net adverse clinical and cerebral events (NACCE) | 1 year
  A composite of all-cause death, any myocardial infarction, stroke, or major bleeding.

SECONDARY OUTCOMES:
All-cause death | 1 year
  All-cause mortality
Any myocardial infarction | 1 year
  According to the Academic Research Consortium (ARC) definition
Stroke | 1 year
  Focal loss of neurologic function caused by an ischemic or hemorrhagic event with residual symptoms lasting at least 24 hours or leading to death
Major Bleeding | 1 year
  Defined by Thrombolysis in Myocardial Infarction (TIMI) major bleeding or TIMI in the setting of coronary artery bypass grafting, and/or any Bleeding Academic Research Consortium (BARC) class 3 or 5.
Any clinically indicated revascularization | 1 year
  Revascularization by PCI or CABG
Stent thrombosis | 1 year
  According to the Academic Research Consortium (ARC) definition

CONTACTS AND LOCATIONS:
Overall Officials: Clemens von Birgelen, MD,PhD,Prof, Study Director — Thoraxcentrum Twente; K. Gert van Houwelingen, MD, Principal Investigator — Thoraxcentrum Twente
Locations (1):
- Medisch Spectrum Twente, Enschede, Netherlands

REFERENCES:
- [Derived] Zocca P, van der Heijden LC, Kok MM, Lowik MM, Hartmann M, Stoel MG, Louwerenburg JW, de Man FHAF, Linssen GCM, Knottnerus IL, Doggen CJM, van Houwelingen KG, von Birgelen C. Clopidogrel or ticagrelor in acute coronary syndrome patients treated with newer-generation drug-eluting stents: CHANGE DAPT. EuroIntervention. 2017 Nov 20;13(10):1168-1176. doi: 10.4244/EIJ-D-17-00634. PMID 29151439